CLINICAL TRIAL: NCT06440564
Title: Laser Disinfection as Biofilm-Disrupter in Periprosthetic Joint Infection (PJI)
Brief Title: Laser Disinfection in Periprosthetic Joint Infection
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Paracelsus Medical University (Other)
Responsible Party: Principal Investigator, Lukas Kriechbaumer, MD, Paracelsus Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1087/2021
Record Dates: First submitted 2024-05-24; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Periprosthetic Joint Infections
Keywords: Er:YAG laser; biofilm removal; periprosthetic joint infections (PJI); DAIR; laser disinfection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Er:YAG Laser intervention (Experimental): In addition to the standard DAIR procedure, laser light is used to disrupt the biofilm from implant surfaced.
  Interventions: Procedure: Er:YAG Laser irradiation

INTERVENTIONS:
Procedure: Er:YAG Laser irradiation — The presented DALIR procedure differs in so far from a standard treatment that after exposure all accessible metal implant surfaces and the adjacent soft tissue is irradiated manually with the Er:YAG laser all over line-by-line with an intended overlap of approximately 10% at constant spot diameter.
  Other Names: Mechanical cleaning with LavaSurge®

SUMMARY:
The eradication of biofilms from infected implants is still an unsolved challenge. The high-energy light beam of an Er:YAG laser causes rapid heating and explosive ablation of tissue. In this study we test the suitability of this laser for the removal of biofilms from infected implant surfaces.

DETAILED DESCRIPTION:
Infections after joint arthroplasties represent a devastating and progressively escalating complication with increased morbidity and mortality. The eradication of biofilms from infected implants is still an unsolved challenge. The high-energy light beam of an Er:YAG laser causes rapid heating and explosive ablation of tissue. In this study the investigators test the suitability of this laser for the removal of biofilms from infected implant surfaces.

Methods In this prospective study, acute or early hematogenous periprosthetic joint infections (PJIs) will be treated with the modified procedure of Debridement, Antibiotics, Laser irradiation and Implant Retention (DALIR). The investigators compare the completeness of biofilm removal from the implant surface with mechanical cleansing alone and the additional use of Er:YAG laser light. Therefore, the investigators will obtain swab cultures from the implants on three distinct occasions: post-arthrotomy, subsequent to mechanical cleansing, and after Er:YAG laser irradiation. The investigators also compare the success rate of the DALIR procedure with the international literature.

Results The investigators expect, that the prevalence of viable microorganisms obtained from implant surfaces through swab cultures will be considerably diminished after additional Er:YAG laser therapy in comparison to only mechanical cleaning with LavaSurge®. The investigators hope to reach a higher healing rate in relation to comparable studies.

Conclusion If the hypothese is correct, the investigators will recommend the use of Er:YAG laser irradiation as an additional tool for disinfection of metal implants in PJIs whenever a DAIR procedure seems to be beneficial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with periprosthetic joint infection (PJI) that will be treated with a debridement, antibiotics, and implant retention (DAIR) procedure

Exclusion Criteria:

* When a DAIR procedure seems not beneficial in a PJI case.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Biofil Eradication | 14 days
  Primary outcome is the comparison of biofilm removal from the implant surface with mechanical cleansing alone (LavaSurge® administered with Pulsavac®) and the additional use of Er:YAG laser light. This is demonstrated by taking microbiological swabs from the implant surface before and after laser treatment.

SECONDARY OUTCOMES:
Healing Rate | 1 year
  Secondary outcome is infection eradication at 1 year following the DALIR procedure. Success of a DALIR procedure will be determined by the absence of antibiotic administration, lack of clinical indications of infection, and absence of infection related subsequent surgical procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Lukas K Kriechbaumer, MD, Principal Investigator — Paracelsus Medical University
Locations (1):
- University Clinic of Orthopedics and Trauma Surgery (Paracelus Medical University Salzburg, Austria), Salzburg, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kriechbaumer LK, Deininger C, Planitzer A, Mitterer M, Happak W, Nurnberger S, Marko P, Filipp S, Thalhammer G, Frenzel S, Hruby L, Korn G. Laser Disinfection Acts as Biofilm-Disrupter in Periprosthetic Joint Infection (PJI). J Orthop Res. 2026 Jan;44(1):e70035. doi: 10.1002/jor.70035. Epub 2025 Jul 23. PMID 40702692